CLINICAL TRIAL: NCT01849653
Title: Self-Obtained Vaginal Swabs for Chlamydia and Gonorrhea Testing: Concurrence in Non-Clinical Settings vs. Clinical Settings
Brief Title: Self-Obtained Vaginal Swabs for Chlamydia and Gonorrhea Testing
Acronym: SOVS-CTG
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: SOVS-CTG2013; HHSN266200400074C (Other Grant/Funding Number: NIH DMID)
Record Dates: First submitted 2013-04-24; First posted 2013-05-08 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Chlamydial Infection; Gonococcal Infection
Keywords: vaginal swabs; diagnosis
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual vaginal swab specimens collected with the APTIMA® Vaginal Swab Specimen Collection Kit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women - Upcoming routine clinic visit: This group of women will self-obtain vaginal swabs at home on the day of their medical appointment and bring the specimens to the clinic. Subjects will then self-obtain another set of vaginal swabs at the clinic. Clinician/nurse will obtain another set of vaginal swabs from the subject at the clinic.
- Women - Recruited while at the clinic: This group of women will self-obtain vaginal swabs at the clinic. Clinician/nurse will obtain another set of vaginal swabs from the subject at the clinic. Within 24 hours of their clinic visit, subjects will self-obtain another set of vaginal swabs at their home and mail them to the laboratory.

SUMMARY:
To evaluate the agreement between NAAT results for Chlamydia trachomatis and Neisseria gonorrhoeae infection obtained with self-obtained vaginal swabs (SOVS), collected in a non-clinical setting vs. NAAT results using SOVS collected in a clinical setting. This is a new use of this specimen type as SOVS are FDA cleared only for use in clinics. The NAAT (Gen-Probe APTIMA Combo 2® Assay (AC2)) result with the home-collected SOVS specimen will be compared to the result obtained with an SOVS collected in the clinic on multiple platforms (Direct Tube Sampling (DTS) / Panther / Tigris). The term "home-collected" is used to refer to any specimen that is not collected in a clinic, since there is no certainty that a specimen is collected "at home" or in a restroom in an office setting, etc. To compare the SOVS results to an FDA cleared predicate test with the collection of two clinician collected vaginal swabs.

DETAILED DESCRIPTION:
All potential participants enrolled in this study will undergo the following procedures:

* Informed consent (written) to participate in this study along with review of the Participant Information Sheet and Experimental Subject's Bill of Rights (per site requirements)
* Assessment of eligibility by nurse/clinician
* Collection of two SOVS in clinic
* Collection of two clinician collected vaginal swabs in the clinic
* Assessment of clinical signs or symptoms
* Group 1 - participants will collect two SOVS before clinic visit and deliver specimens to study staff at the clinic visit.
* Group 2 - participants will repeat collection of two SOVS at home after clinic visit and mail the specimens directly to the laboratory.

Clinical examinations will be conducted as appropriate to the reason for the visit/exam but the clinic procedures are not included as part of the protocol.

The enrollment strategy is designed to recruit a total of 3500 women with an average of 42-60 women per month over a 12-month recruitment period (500-700 women per site over the recruitment period). Participants will be seen and recruited in clinics at the participating STI-CTG, and other site clinics. At each participating clinical center, recruitment personnel will follow a site specific process that is designed to help identify potential participants. Only one visit is required to complete the study procedures. The total time required for a participant to complete this study may vary but is expected to be 45 minutes total time over 1 or 2 days. Intervals of several days between collection of the two specimens are likely for some women.

Clinic staff will approach women in the clinic or via phone and explain the object of the study and requirements of participation. The consenting process adopted by each site will be dependent on their IRB approval. Written consent will be obtained for all participants.

Participants will be given a Participant Information Sheet to read and keep. [In addition, sites and clinics in California must utilize the "Experimental Subject's Bill of Rights" that explains their rights as a research subject per California law.] For Group 1, the discussions will be by phone and the Information Sheet and Experimental Subject's Bill of Rights will be included in the collection kit that is mailed to participants. Clinic staff will utilize a standard script including a form of Q&A to ensure that participants have a basic understanding of the SOVS procedures. Participants will be encouraged to call the clinic staff with any questions when they receive the home collection kit.

After the participant provides informed consent, the nurse/clinician will assign a unique participant number (PN) and note the consenting procedure and appropriate eligibility information on a Case Report Form (CRF). The nurse/clinician will discuss basic demographic, medical history and concomitant medication information with each participant and record the information either on a study specific notes page, or a CRF. These will be maintained in the participant's research study record. This information will be used to assess eligibility. Participants in both study groups will be provided with swab collection kits along with a diagram showing how to collect the SOVS specimens. The participant will collect the swabs in a designated place in the clinic (often a rest room) at the beginning of the visit before any other specimens are collected. Next, the nurse/clinician will conduct the examination to manage the participant's healthcare. If the standard of care at the clinic is an SOVS processed using AC2, the participant will undergo an additional specimen collection as per the local clinic's standard of care for diagnosis and management of Ct/GC. Standard protocols for clinical management may differ by study site and will not be modified as a result of this study. Beyond the laboratory's AC2 Ct/GC NAAT clinical results, site standard protocols are not relevant to this study. Participants will not be notified regarding test results from the SOVS collected solely for this study. This will end the Study participation for Group 1.

At the end of the clinic visit for Group 2 participants, the nurse/clinician will provide them with the HOLOGIC|Gen-Probe, Inc. provided home swab collection kits (the same as those mailed to participants in Group 1). The kits are identical to the kits used in the clinic with the addition of a mailing container and relevant mailing labels. Participants will be instructed to return home (or to another non-clinical private location) and collect two additional specimens:

* within 24 hours of the clinic visit
* prior to resuming sexual activity
* prior to taking any antibiotics that have been prescribed

Group 2 participants will then mail the specimens to the laboratory in the mailer provided within 24 hours of collecting the sample. Participants will be given the same instructions for collecting the swabs regardless of whether it is in the clinic restroom or at home. Group 2 participants will receive a follow-up communication 48 hours after their clinic appointment.

Participants in both groups will complete all other study procedures at the clinic during the initial visit. One questionnaire will be administered to the participants (the Home-collected SOVS CRF) and only the following clinical data will be collected as part of this study - participant's age, gender, race/ethnicity, clinical signs & symptoms, date of exam, date/time specimen collected/mailed/received, UADEs (if any), and AC2 results.

All laboratory evaluations will use the APTIMA Combo 2® assay for detection of Ct/GC infection on the SOVS specimens collected "at home" and "in clinic" across 3 different platforms (DTS, Panther, and Tigris). One set of specimen collection tubes ("at home" and "in clinic") will be tested on DTS at each of 5 to 7 laboratories associated with the clinical sites. A matched set of specimen collection tubes will be shipped to 1 of 3 designated laboratory sites to be tested on Panther. Once the Panther testing is completed, the same set of tubes will be shipped to 1 of 3 different laboratory sites to be tested on Tigris. Results will be compared to assess agreement of the paired specimens tested within each platform (DTS / Panther / Tigris).

The APTIMA Combo 2® Assay (HOLOGIC | Gen-Probe Inc., San Diego, CA) is a nucleic acid amplification test (NAAT) that utilizes target capture for the detection and differentiation of ribosomal RNA (rRNA) from Chlamydia trachomatis and/or Neisseria gonorrhoeae in clinician-collected endocervical, vaginal (VS-C), and male urethral swab specimens, SOVS specimens (when obtained in the clinic), and female and male urine specimens. The assay is FDA cleared for use with specimens from symptomatic and asymptomatic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic and symptomatic females ages 16-75
* Subjects scheduled for visits or presenting at Family Planning, OB/Gyn, STD or other clinics requesting (or candidates for) routine screening for Ct/GC
* Willing to provide informed consent (written per site institutional review board approval)

Exclusion Criteria:

* Inability to provide informed consent
* Inability or unwillingness to collect a specimen at home (and mail it)
* On antibiotic therapy within the last 30 days
* Clinical conditions, such as cervicitis or pelvic inflammatory disease that would indicate presumptive treatment
* Contact to person with Ct or GC in need of epidemiologic treatment

Ages: 16 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This will be a multicenter trial involving approximately 3500 women ages 16-75 from different geographic areas in North America and from populations having different prevalences of Ct and GC. Women will be either healthy women having routine exams, or women being evaluated specifically for STDs (symptomatic and asymptomatic). Sites will include Family Planning, Ob/Gyn and STD clinics. The possibility of using a college student health clinic and a military clinic will be explored if it proves feasible to obtain a large enough number of participants during the project's planned duration.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Chlamydia trachomatis detected by nucleic acid amplification test in vaginal swabs | 24 hrs (at clinic visit)
  AC2 testing on the DTS, Panther, and Tigris platforms for the presence or absence of Ct on "Home-collected" vs. "Clinic-collected" swab specimens, and clinician collected swabs.

SECONDARY OUTCOMES:
Neisseria gonorrhoeae detected by nucleic acid amplification test in vaginal swabs | 24 hrs (at clinic visit)
  AC2 testing on the DTS, Panther, and Tigris platforms for the presence or absence of GC on "Home-collected" vs. "Clinic-collected" swab specimens, and clinician collected swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Julius Schachter, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Hobbs MM, van der Pol B, Totten P, Gaydos CA, Wald A, Warren T, Winer RL, Cook RL, Deal CD, Rogers ME, Schachter J, Holmes KK, Martin DH. From the NIH: proceedings of a workshop on the importance of self-obtained vaginal specimens for detection of sexually transmitted infections. Sex Transm Dis. 2008 Jan;35(1):8-13. doi: 10.1097/OLQ.0b013e31815d968d. PMID 18157061
- [Background] Martin DH, Cammarata C. Potential causes of decreased sensitivity of the Abbott ligase chain reaction (LCR) assay for Chlamydia trachomatis (Ct) in urine specimens. 13th International Society for Sexually Transmitted Diseases Research (ISSTDR). Denver, CO; 1999.
- [Background] Kudrick JA, (DMID Clinical Agents Repository Contract: Fisher BioServices). Personal correspondence with NIH/NIAID staff. Germantown, MD; February 10, 2011.
- [Background] Altman DG, Machin D, Bryant TN, Gardner MJ, (eds). Statistics with Confidence, 2nd ed. Bristol, UK: British Medical Journal; 2000.
- [Background] Shafer MA, Pantell RH, Schachter J. Is the routine pelvic examination needed with the advent of urine-based screening for sexually transmitted diseases? Arch Pediatr Adolesc Med. 1999 Feb;153(2):119-25. doi: 10.1001/archpedi.153.2.119. PMID 9988241
- [Result] Xu F, Stoner BP, Taylor SN, Mena L, Tian LH, Papp J, Hutchins K, Martin DH, Markowitz LE. Use of home-obtained vaginal swabs to facilitate rescreening for Chlamydia trachomatis infections: two randomized controlled trials. Obstet Gynecol. 2011 Aug;118(2 Pt 1):231-239. doi: 10.1097/AOG.0b013e3182246a83. PMID 21775837
- [Result] Gotz HM, van den Broek IV, Hoebe CJ, Brouwers EE, Pars LL, Fennema JS, Koekenbier RH, van Ravesteijn S, Op de Coul EL, van Bergen J. High yield of reinfections by home-based automatic rescreening of Chlamydia positives in a large-scale register-based screening programme and determinants of repeat infections. Sex Transm Infect. 2013 Feb;89(1):63-9. doi: 10.1136/sextrans-2011-050455. Epub 2012 Jun 23. PMID 22728910
- [Result] Cook RL, Ostergaard L, Hillier SL, Murray PJ, Chang CC, Comer DM, Ness RB; DAISY study team. Home screening for sexually transmitted diseases in high-risk young women: randomised controlled trial. Sex Transm Infect. 2007 Jul;83(4):286-91. doi: 10.1136/sti.2006.023762. Epub 2007 Feb 14. PMID 17301105
- [Result] Gaydos CA, Barnes M, Aumakhan B, Quinn N, Wright C, Agreda P, Whittle P, Hogan T. Chlamydia trachomatis age-specific prevalence in women who used an internet-based self-screening program compared to women who were screened in family planning clinics. Sex Transm Dis. 2011 Feb;38(2):74-8. doi: 10.1097/OLQ.0b013e3182039d7f. PMID 21173720
- [Result] Schachter J, Chow JM, Howard H, Bolan G, Moncada J. Detection of Chlamydia trachomatis by nucleic acid amplification testing: our evaluation suggests that CDC-recommended approaches for confirmatory testing are ill-advised. J Clin Microbiol. 2006 Jul;44(7):2512-7. doi: 10.1128/JCM.02620-05. PMID 16825373
- [Result] Lee HH, Chernesky MA, Schachter J, Burczak JD, Andrews WW, Muldoon S, Leckie G, Stamm WE. Diagnosis of Chlamydia trachomatis genitourinary infection in women by ligase chain reaction assay of urine. Lancet. 1995 Jan 28;345(8944):213-6. doi: 10.1016/s0140-6736(95)90221-x. PMID 7823713
- [Result] Hook EW 3rd, Smith K, Mullen C, Stephens J, Rinehardt L, Pate MS, Lee HH. Diagnosis of genitourinary Chlamydia trachomatis infections by using the ligase chain reaction on patient-obtained vaginal swabs. J Clin Microbiol. 1997 Aug;35(8):2133-5. doi: 10.1128/jcm.35.8.2133-2135.1997. PMID 9230397
- [Result] Stary A, Najim B, Lee HH. Vulval swabs as alternative specimens for ligase chain reaction detection of genital chlamydial infection in women. J Clin Microbiol. 1997 Apr;35(4):836-8. doi: 10.1128/jcm.35.4.836-838.1997. PMID 9157137
- [Result] Schachter J, McCormack WM, Chernesky MA, Martin DH, Van Der Pol B, Rice PA, Hook EW 3rd, Stamm WE, Quinn TC, Chow JM. Vaginal swabs are appropriate specimens for diagnosis of genital tract infection with Chlamydia trachomatis. J Clin Microbiol. 2003 Aug;41(8):3784-9. doi: 10.1128/JCM.41.8.3784-3789.2003. PMID 12904390
- [Result] Schachter J, Chernesky MA, Willis DE, Fine PM, Martin DH, Fuller D, Jordan JA, Janda W, Hook EW 3rd. Vaginal swabs are the specimens of choice when screening for Chlamydia trachomatis and Neisseria gonorrhoeae: results from a multicenter evaluation of the APTIMA assays for both infections. Sex Transm Dis. 2005 Dec;32(12):725-8. doi: 10.1097/01.olq.0000190092.59482.96. PMID 16314767
- [Result] Chernesky MA, Hook EW 3rd, Martin DH, Lane J, Johnson R, Jordan JA, Fuller D, Willis DE, Fine PM, Janda WM, Schachter J. Women find it easy and prefer to collect their own vaginal swabs to diagnose Chlamydia trachomatis or Neisseria gonorrhoeae infections. Sex Transm Dis. 2005 Dec;32(12):729-33. doi: 10.1097/01.olq.0000190057.61633.8d. PMID 16314768
- [Result] Shafer MA, Moncada J, Boyer CB, Betsinger K, Flinn SD, Schachter J. Comparing first-void urine specimens, self-collected vaginal swabs, and endocervical specimens to detect Chlamydia trachomatis and Neisseria gonorrhoeae by a nucleic acid amplification test. J Clin Microbiol. 2003 Sep;41(9):4395-9. doi: 10.1128/JCM.41.9.4395-4399.2003. PMID 12958275
- [Result] Macmillan S, McKenzie H, Templeton A. Parallel observation of four methods for screening women under 25 years of age for genital infection with Chlamydia trachomatis. Eur J Obstet Gynecol Reprod Biol. 2003 Mar 26;107(1):68-73. doi: 10.1016/s0301-2115(02)00266-x. PMID 12593898
- [Result] Oakeshott P, Hay P, Hay S, Steinke F, Rink E, Thomas B, Oakeley P, Kerry S. Detection of Chlamydia trachomatis infection in early pregnancy using self-administered vaginal swabs and first pass urines: a cross-sectional community-based survey. Br J Gen Pract. 2002 Oct;52(483):830-2. PMID 12392124
- [Result] Smith K, Harrington K, Wingood G, Oh MK, Hook EW 3rd, DiClemente RJ. Self-obtained vaginal swabs for diagnosis of treatable sexually transmitted diseases in adolescent girls. Arch Pediatr Adolesc Med. 2001 Jun;155(6):676-9. doi: 10.1001/archpedi.155.6.676. PMID 11386956
- [Result] Gaydos CA, Crotchfelt KA, Shah N, Tennant M, Quinn TC, Gaydos JC, McKee KT Jr, Rompalo AM. Evaluation of dry and wet transported intravaginal swabs in detection of Chlamydia trachomatis and Neisseria gonorrhoeae infections in female soldiers by PCR. J Clin Microbiol. 2002 Mar;40(3):758-61. doi: 10.1128/JCM.40.3.758-761.2002. PMID 11880389
- [Result] Chernesky M, Jang D, Luinstra K, Chong S, Smieja M, Cai W, Hayhoe B, Portillo E, Macritchie C, Main C, Ewert R. High analytical sensitivity and low rates of inhibition may contribute to detection of Chlamydia trachomatis in significantly more women by the APTIMA Combo 2 assay. J Clin Microbiol. 2006 Feb;44(2):400-5. doi: 10.1128/JCM.44.2.400-405.2006. PMID 16455891
- See also: Association of Public Health Laboratories (APHL). Laboratory Diagnostic Testing for Chlamydia trachomatis and Neisseria gonorrhoeae. Expert Consultation Meeting Summary Report, January 13-15, 2009 — http://www.aphl.org/aphlprograms/infectious/std/Documents/ID_2009Jan_CTGCLab-Guidelines-Meeting-Report.pdf